CLINICAL TRIAL: NCT02479139
Title: Clinical Trial to Evaluate ANT-1207 in the Treatment of Primary Axillary Hyperhidrosis in Adults
Brief Title: Clinical Trial To Evaluate ANT-1207 In Participants With Primary Axillary Hyperhidrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANT-1207-HHID-205
Record Dates: First submitted 2015-06-19; First posted 2015-06-24 (Estimated); Results first posted 2017-09-20 (Actual); Last update posted 2017-09-20 (Actual); Status verified 2017-08

CONDITIONS: Hyperhidrosis
MeSH Terms: conditions — Hyperhidrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Vehicle (Placebo Comparator): Vehicle for botulinum toxin Type A topical liniment (ANT-1207) applied topically in a volume of 12 drops per axilla (armpit) once on Day 0.
  Interventions: Biological: Vehicle
- ANT-1207 Dose 1 (Experimental): Botulinum toxin Type A topical liniment (ANT-1207) Dose 1 (lowest dose) applied topically in a volume of 12 drops per axilla (armpit) once on Day 0.
  Interventions: Biological: ANT-1207
- ANT-1207 Dose 2 (Experimental): Botulinum toxin Type A topical liniment (ANT-1207) Dose 2 (second lowest dose) applied topically in a volume of 12 drops per axilla (armpit) once on Day 0.
  Interventions: Biological: ANT-1207
- ANT-1207 Dose 3 (Experimental): Botulinum toxin Type A topical liniment (ANT-1207) Dose 3 (mid-level dose) applied topically in a volume of 12 drops per axilla (armpit) once on Day 0.
  Interventions: Biological: ANT-1207
- ANT-1207 Dose 4 (Experimental): Botulinum toxin Type A topical liniment (ANT-1207) Dose 4 (second highest dose) applied topically in a volume of 12 drops per axilla (armpit) once on Day 0.
  Interventions: Biological: ANT-1207
- ANT-1207 Dose 5 (Experimental): Botulinum toxin Type A topical liniment (ANT-1207) Dose 5 (highest dose) applied topically in a volume of 12 drops per axilla (armpit) once on Day 0.
  Interventions: Biological: ANT-1207

INTERVENTIONS:
Biological: Vehicle — Vehicle for ANT-1207 liniment formulation without active ingredient.
  Arms: Vehicle
Biological: ANT-1207 — Botulinum toxin Type A topical liniment (ANT-1207).
  Arms: ANT-1207 Dose 1; ANT-1207 Dose 2; ANT-1207 Dose 3; ANT-1207 Dose 4; ANT-1207 Dose 5

SUMMARY:
The purpose of this study is to establish the therapeutic range of ANT-1207 in the treatment of primary axillary hyperhidrosis.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 - 70 years of age
* diagnosis of primary axillary hyperhidrosis
* HDSS score of ≥3
* threshold sweat production/axilla in 5 minutes as measured gravimetrically
* willingness to shave underarms prior to each study visit

Exclusion Criteria:

* botulinum toxin treatment in the prior 6 months
* signs of infection in the axilla
* skin affliction in the axilla requiring medical treatment
* oral anticholinergic treatment
* use of antiperspirants, deodorants, powders, or lotions
* use of axillary depilatories or axillary epilation
* history of surgery or other interventions for axillary hyperhidrosis
* female subjects who are pregnant or are nursing a child

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2015-06-03 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan-En Lin, Study Director — Allergan
Locations (19):
- United States (19):
  - San Marcus Research Clinic, Inc., Hialeah, Florida
  - Baumann Cosmetic & Research Institute, Miami, Florida
  - Radiant Research, Inc., Pinellas Park, Florida
  - Research Institute of the Southeast, LLC, West Palm Beach, Florida
  - Shideler Clinical Research Center, Carmel, Indiana
  - William Coleman III, MD, APMC, Metairie, Louisiana
  - Lupo Center for Aesthetic & General Dermatology, New Orleans, Louisiana
  - Skin Specialists, PC, Omaha, Nebraska
  - JUVA Skin and Laser Center, New York, New York
  - Skin Search of Rochester, Inc., Rochester, New York
  - PMG Research of Cary, Cary, North Carolina
  - Allus Clinical Research, Jenkintown, Pennsylvania
  - Dermatology and Laser Center of Charleston, PA, Charleston, South Carolina
  - The Skin Wellness Center, Knoxville, Tennessee
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - J&S Studies, Inc., College Station, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research Inc., Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vehicle | ANT-1207 Dose 1 | ANT-1207 Dose 2 | ANT-1207 Dose 3 | ANT-1207 Dose 4 | ANT-1207 Dose 5
Started | 27 | 22 | 28 | 21 | 22 | 25
Completed | 19 | 12 | 21 | 14 | 17 | 19
Not Completed | 8 | 10 | 7 | 7 | 5 | 6
Not completed — Lost to Follow-up | 2 | 4 | 4 | 2 | 3 | 5
Not completed — Withdrew Consent | 5 | 6 | 1 | 4 | 1 | 1
Not completed — Treatment Failure/Lack of Efficacy | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Other Miscellaneous Reasons | 1 | 0 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vehicle | ANT-1207 Dose 1 | ANT-1207 Dose 2 | ANT-1207 Dose 3 | ANT-1207 Dose 4 | ANT-1207 Dose 5 | Total
Number analyzed (Participants) | 27 | 22 | 28 | 21 | 22 | 25 | 145
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.15 (11.83) | 30.18 (6.70) | 32.50 (9.86) | 30.48 (6.90) | 32.36 (9.56) | 32.64 (10.55) | 31.79 (9.46)
Age, Customized [Number; unit: participants]
  18 to 35 years | 19 | 18 | 19 | 16 | 13 | 17 | 102
  36 to 50 years | 5 | 4 | 8 | 5 | 8 | 7 | 37
  >50 years | 3 | 0 | 1 | 0 | 1 | 1 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 12 | 17 | 14 | 11 | 12 | 82
  Male | 11 | 10 | 11 | 07 | 11 | 13 | 63

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Both a Change From Baseline in Hyperhidrosis Disease Severity Scale (HDSS) Score by ≥ 2 Points and a Change From Baseline in Gravimetric Sweat Production (GSP) by ≥ 50%
Description: The HDSS is a patient completed scale that measures how excessive sweating effects quality of life using a 4-point scale where: 1=My underarm sweating is not noticeable and never interferes with my daily activities to 4= My underarm sweating is intolerable and always interferes with my daily activities.
  GSP was measured using a pre-weighed filter paper placed into the axilla area (armpit) to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced.
  The HDSS and the GSP were assessed at Baseline and Week 12. The change from Baseline was calculated. The percentage of participants who had both a change (reduction) from Baseline in HDSS score by ≥ 2 points and a change (reduction) from Baseline in GSP by ≥ 50% is reported.
Time Frame: Baseline, Week 12
Population: Modified Intent-to-Treat (mITT) population was defined as all randomized participants who received at least 1 dose of investigational product with both a baseline value and ≥ 1 value during the double-blind treatment period. Missing values were imputed using the last observation carried forward (LOCF) approach.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | ANT-1207 Dose 1 | ANT-1207 Dose 2 | ANT-1207 Dose 3 | ANT-1207 Dose 4 | ANT-1207 Dose 5
Number analyzed (Participants) | 27 | 22 | 28 | 21 | 21 | 25
percentage of participants | 3.70 | 13.64 | 17.86 | 14.29 | 14.29 | 12.00

2. Secondary Outcome: Percentage of Participants With Hyperhidrosis Disease Severity Scale (HDSS) Score Change From Baseline ≥ 2 Points
Description: The HDSS is a patient completed scale that measures how excessive sweating effects quality of life using a 4-point scale where: 1=My underarm sweating is not noticeable and never interferes with my daily activities to 4= My underarm sweating is intolerable and always interferes with my daily activities.
  The change from Baseline was calculated. The percentage of participants who had a change (reduction) from Baseline in HDSS score by ≥ 2 points is reported.
Time Frame: Baseline, Weeks 4, 8, 12 and 18
Population: mITT population was defined as all randomized participants who received at least 1 dose of investigational product with both a baseline value and ≥ 1 value during the double-blind treatment period. Missing values were imputed using the LOCF approach.
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | ANT-1207 Dose 1 | ANT-1207 Dose 2 | ANT-1207 Dose 3 | ANT-1207 Dose 4 | ANT-1207 Dose 5
Number analyzed (Participants) | 27 | 22 | 28 | 21 | 21 | 25
percentage of participants
  Week 4 | 29.63 | 13.64 | 21.43 | 9.52 | 28.57 | 16.00
  Week 8 | 11.11 | 22.73 | 28.57 | 19.05 | 14.29 | 4.00
  Week 12 | 7.41 | 27.27 | 25.00 | 19.05 | 14.29 | 12.00
  Week 18 | 7.41 | 22.73 | 21.43 | 19.05 | 23.81 | 8.00

3. Secondary Outcome: Percentage of Participants With Gravimetric Sweat Production (GSP) Change From Baseline ≥ 50%
Description: GSP was measured using a pre-weighed filter paper placed into the axilla area (armpit) to collect sweat over a 5-minute period. The paper was removed and weighed to determine the amount of sweat produced.
  The change from Baseline was calculated. The percentage of participants who had a change (reduction) from Baseline in GSP by ≥ 50% is reported.
Time Frame: Baseline, Weeks 4, 8, 12 and 18
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Vehicle | ANT-1207 Dose 1 | ANT-1207 Dose 2 | ANT-1207 Dose 3 | ANT-1207 Dose 4 | ANT-1207 Dose 5
Number analyzed (Participants) | 27 | 22 | 28 | 21 | 21 | 25
percentage of participants
  Week 4 | 62.96 | 72.73 | 71.43 | 71.43 | 61.90 | 72.00
  Week 8 | 55.56 | 72.73 | 71.43 | 57.14 | 52.38 | 72.00
  Week 12 | 66.67 | 63.64 | 67.86 | 47.62 | 71.43 | 72.00
  Week 18 | 51.85 | 54.55 | 64.29 | 47.62 | 61.90 | 76.00

ADVERSE EVENTS:
Time Frame: 126 Days
Description: Safety population included all randomized patients who received at least 1 dose of double-blind investigational product.
Arm/Group | Vehicle | ANT-1207 Dose 1 | ANT-1207 Dose 2 | ANT-1207 Dose 3 | ANT-1207 Dose 4 | ANT-1207 Dose 5
Serious Adverse Events (participants affected / at risk) | 1/27 | 0/22 | 0/28 | 0/21 | 0/22 | 0/25
Other Adverse Events (participants affected / at risk) | 0/27 | 0/22 | 2/28 | 0/21 | 0/22 | 1/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=27) | ANT-1207 Dose 1 (N=22) | ANT-1207 Dose 2 (N=28) | ANT-1207 Dose 3 (N=21) | ANT-1207 Dose 4 (N=22) | ANT-1207 Dose 5 (N=25)
Gastrectomy (Surgical and medical procedures) | 1 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vehicle (N=27) | ANT-1207 Dose 1 (N=22) | ANT-1207 Dose 2 (N=28) | ANT-1207 Dose 3 (N=21) | ANT-1207 Dose 4 (N=22) | ANT-1207 Dose 5 (N=25)
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.